CLINICAL TRIAL: NCT03561311
Title: The Neuroprotective Effect of Remote Ischemic Conditioning in Ruptured Aneurysm Coiling Therapy
Acronym: NEAT-2
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Principal Investigator, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-NEAT-2
Record Dates: First submitted 2018-05-23; First posted 2018-06-19 (Actual); Last update posted 2018-11-23 (Actual); Status verified 2018-11

CONDITIONS: Aneurysm, Ruptured; Coiling Therapy
MeSH Terms: conditions — Aneurysm, Ruptured

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remote ischemic conditioning group (Experimental)
  Interventions: Device: remote ischemic conditioning
- Sham remote ischemic conditioning group (Sham Comparator)
  Interventions: Device: sham remote ischemic conditioning

INTERVENTIONS:
Device: remote ischemic conditioning — Remote ischemic conditioning is performed by using an electric autocontrol device with cuffs that inflated to a pressure of 200 mm Hg during the ischemic period (Patent No. CN200820123637.X, China)
  Arms: Remote ischemic conditioning group
Device: sham remote ischemic conditioning — Sham remote ischemic conditioning is performed by using an electric autocontrol device with cuffs that inflated to a pressure of 60 mm Hg
  Arms: Sham remote ischemic conditioning group

SUMMARY:
The overall incidence of DWI positive for thromboembolic events following endovascular treatment of intracranial aneurysms is proximately 50%. Whether remote ischemic conditioning was safe and effective to reduce ischemic brain lesions on DWI after endovascular treatment of intracranial aneurysms is still unclear. The investigators' hypothesis is that remote ischemic conditioning is a safe and effective strategy to reduce new ischemic lesions in intracranial aneurysms patients undergoing endovascular treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Ruptured brain aneurysm deemed suitable for neuroendovascular repair
* Normal baseline brain MRI
* Female subjects of childbearing potential have a negative pregnancy test.
* Signed informed consent prior to entering study

Exclusion Criteria:

* Dissecting or mycotic brain aneurysm.
* Planned endovascular vessel sacrifice as the primary modality for aneurysm treatment
* Renal insufficiency with creatinine ≥ 265 umol/L
* Severe, sustained hypertension (SBP > 185 mmHg or DBP > 110 mmHg)
* Contraindication for remote ischemic conditioning: severe soft tissue injury, fracture, or peripheral vascular disease in the upper limbs
* Pre-morbid modified Rankin scale score of greater than 1
* Patients with a pre-existing neurological or psychiatric disease that would confound the neurological or functional evaluations Patients who are unable to have an MRI scan for any reason.
* Currently participating or previously participated in any investigational drug or device study within 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2018-10-06 (Actual); Primary Completion 2019-05-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
The presence of ≥1 new brain lesions on DWI | within 72 hours after endovascular treatment
  Assessed by DWI

SECONDARY OUTCOMES:
Number of new ischemic lesions | within 72 hours after endovascular treatment
Volume of new ischemic lesions | within 72 hours after endovascular treatment
National Institutes of Health Stroke Scale | 7 days or discharge
  Scores on the National Institutes of Health Stroke Scale (NIHSS) range from 0 to 42, with higher scores indicating more severe neurologic deficits.
Composite of Cerebrovascular events | 30 days
  This is a composited endpoint.Cerebrovascular events included ischemic stroke, hemorrhagic stroke, and TIA. The present subarachnoid hemorrhage isn't included.
Nondisabling events | 30 days
  Scores on the National Institutes of Health Stroke Scale (NIHSS) range from 0 to 42, with higher scores indicating more severe neurologic deficits.National Institutes of Health Stroke Scale ≤3 or TIA is defined as nondisabling events The present subarachnoid hemorrhage isn't included.
Modified Rankin Scale | 30 days
  Scores on the modified Rankin scale of functional disability range from 0 (no symptoms) to 6 (death).

OTHER OUTCOMES:
Occurrence of adverse events and serious adverse events | 30 days
  Occurrence of adverse events and serious adverse events

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Shengli Oilfield Central Hospital, Dongying, Shandong
  - The Second People's Hospital of Liaocheng, Liaocheng
  - Nanyang City Center Hospital, Nanyang
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou